CLINICAL TRIAL: NCT00261196
Title: Collagenase in the Treatment of Adhesive Capsulitis (Frozen Shoulder)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IND moved to sponsor.
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Marie Badalamente, Professor Orthopaedics, Stony Brook University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Shoulder 202
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Adhesive Capsulitis; Frozen Shoulder
Keywords: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Collagenases; Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase (Experimental): Collagenase Injection
  Interventions: Drug: Collagenase
- Placebo (Placebo Comparator): Placebo Injection
  Interventions: Drug: Collagenase

INTERVENTIONS:
Drug: Collagenase — Anterior shoulder capsule injection
  Other Names: Xiaflex

SUMMARY:
The purpose of this study is to test collagenase injection therapy to dissolve adhesions causing frozen shoulder.

DETAILED DESCRIPTION:
In a random, placebo controlled, double blind study, collagenase injection therapy will be investigated for it's ability to lyse the adhesions associated with the shoulder capsule in adhesive capsulitis (frozen shoulder).

Treatment success may obviate the need for extensive physical therapy and/or shoulder arthroscopy (surgery) to correct this condition and restore normal and pain free shoulder motion.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of frozen shoulder of at least one month duration

Exclusion Criteria:

* shoulder arthritis
* rotator cuff tears
* any chronic, serious, uncontrolled medical condition
* inability to conform to study visits (20-30 per year)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Active elevation of the affected shoulder | 30 days
  Active Elevation in degrees by goniometer measurement

SECONDARY OUTCOMES:
Active and passive shoulder motions in internal/external rotation, passive elevation, pain and function. | 30 days
  Active and passive internal/external rotation in degrees by goniometer measure

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Badalamente, PhD, Principal Investigator — Dept. Orthopaedics, SUNY@Stony Brook, NY 11794
Locations (1):
- Dept. Orthopaedics, SUNY@Stony Brook, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No